CLINICAL TRIAL: NCT04774640
Title: Noninvasive In Vitro Diagnostic Test For Fetal Chromosomal Abnormality: Assay Development and Optimization in Affected Pregnancies With Abnormal Microarray Findings
Brief Title: Development of a NIPTT for Detecting Copy Number Variations
Status: Terminated | Type: Observational
Why Stopped: Poor rate of eligible subject enrollment
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: SQNM-T21-306
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2021-02

CONDITIONS: Copy Number Variations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal plasma with cell free fetal DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MaterniT GENOME

SUMMARY:
To collect whole blood samples from pregnant women for the purpose of developing, optimizing and evaluating laboratory-developed noninvasive prenatal test (NIPT) for the detection of fetal chromosomal abnormalities of interest defined as microinsertions, microdeletions and other copy number variations (CNVs). The NIPT result will be compared to the test results obtained by microarray analysis of fetal cellular material obtained by amniocentesis or chorionic villus sampling.

DETAILED DESCRIPTION:
This is a single center specimen collection study. Eligible subjects from across the USA will be referred to the single center for participation.

This study will evaluate whether the test methods being developed for the detection of fetal chromosomal abnormalities of interest in maternal whole blood samples can be used in clinical practice.

Enrollment of study subjects will be done in two phases - an initial pilot study phase to collect samples for research and development activities, followed by a larger single-blinded sample collection phase for NIPT evaluation. For both phases, study subjects will be enrolled in a prospective manner until the predetermined sample size is attained. Each study subject will be asked to provide one 20mL blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female
* Subject is 18 years of age or older
* Subject is pregnant at no less than 10 weeks and no more than 36 weeks gestation
* Subject provides a signed and dated informed consent
* Subject has a current pregnancy in which the fetus is determined to have a chormosomal abnormality of interest (microinsertions, microdeletions and other CNVs) as determined by microarray analysis of fetal cellular material obtained by IP

Exclusion Criteria:

* Subject has experienced fetal demise in the current pregnancy

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects must be pregnant
Study Population: Pregnant women with a fetus previously determined by microarray to have a chromosomal abnormality of interest..
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Development of non-invasive pregnancy test (NIPT) | 5 years
  NIPT results will be compared to test results obtain by microarray analysis of fetal cellular material obtained by amniocentesis or chorionic villus sampling

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No